CLINICAL TRIAL: NCT00213811
Title: Bardet-Biedl Syndrome: Clinical and Genetic Epidemiology Study in the Adults
Brief Title: Bardet-Biedl Syndrome Study: Clinical and Genetic Epidemiology Study in Adults
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Other Study IDs: 2899
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2008-08-08 (Estimated); Status verified 2008-08

CONDITIONS: Bardet-Biedl Syndrome; Orphan Diseases
Keywords: Bardet-Biedl syndrome, retinitis pigmentosa, obesity, genes
MeSH Terms: conditions — Bardet-Biedl Syndrome; Rare Diseases; Retinitis Pigmentosa; Obesity | interventions — Biological Products

INTERVENTIONS:
Behavioral: clinical, biological, and radiological

SUMMARY:
This study is based on the study of the natural history of a rare disorder: the Bardet-Biedl syndrome (BBS) (which is associated with retinitis pigmentosa, polydactyly, cognitive impairment, obesity, and kidney failure). The clinical, biological, and radiological features of adult patients are studied. In parallel, a molecular study is performed on the known genes to date (8 genes from BBS1 to BBS8) and to identify new genes involved. The parts of the study are combined in a phenotype-genotype correlation study.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age over 16 years old)
* At least 3 of the five major criteria (retinitis pigmentosa, obesity, polydactyly, cognitive impairment, and kidney disorder) and/or BBS mutations identified

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2003-06

PRIMARY OUTCOMES:
Outcome evaluated end 2005 and 2006
Clinical results (natural history, phenotype-genotype correlations, genetic epidemiology, new genes identification

SECONDARY OUTCOMES:
This study may lead to further clinical investigations according to the results (new protocol to be established) and to further molecular investigations

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Dollfus, MD, Principal Investigator — Fédération Génétique; J-Louis Mandel, MD, Principal Investigator — IGBMC; Pascal Bousquet, MD, Principal Investigator — CIC Strasbourg; Christian Brandt, MD, Principal Investigator — CIC Strasbourg; Catherine Arnold, MD, Principal Investigator — CIC Strasbourg; Alain Verloes, MD, Principal Investigator — Unité de Génétique Robert Debré; Régis Hanfard, MD, Principal Investigator — CIC Robet Debré; Didier Lacombe, MD, Principal Investigator — Service de Génétique Médicale/Bordeaux; Virginie Bernard, MD, Principal Investigator — CIC Bordeaux; Sylvie Manouvrier, MD, Principal Investigator — Service de Génétique Médicale Lille
Locations (1):
- Hélène Dollfus, Strasbourg, France